CLINICAL TRIAL: NCT02426372
Title: An Open Label, Dose Ranging, Exploratory Study to Evaluate the Safety, Tolerability, Compliance, Mechanism of Action and Efficacy of QBECO Site Specific Immunomodulation for the Induction of Clinical Response and Remission in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Safety and Efficacy of QBECO in Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qu Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QBECO-UC-01
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QBECO SSI 0.02 mL (Experimental): 0.02 mL administered subcutaneously, every other day for 16 weeks. After completion of the initial 16-week fixed dose treatment period, subjects deemed to be responders will be randomized to one of three maintenance dosing schedules (every second day, weekly, no treatment) for an additional 36 weeks.
  Interventions: Biological: QBECO SSI
- QBECO SSI 0.05 mL (Experimental): 0.05 mL administered subcutaneously, every other day for 16 weeks. After completion of the initial 16-week fixed dose treatment period, subjects deemed to be responders will be randomized to one of three maintenance dosing schedules (every second day, weekly, no treatment) for an additional 36 weeks.
  Interventions: Biological: QBECO SSI
- QBECO SSI 0.1 mL (Experimental): 0.1 mL administered subcutaneously, every other day for 16 weeks. After completion of the initial 16-week fixed dose treatment period, subjects deemed to be responders will be randomized to one of three maintenance dosing schedules (every second day, weekly, no treatment) for an additional 36 weeks.
  Interventions: Biological: QBECO SSI

INTERVENTIONS:
Biological: QBECO SSI — QBECO Site Specific Immunomodulators

SUMMARY:
The purpose of this open-label, dose-ranging, exploratory study is to evaluate the safety, tolerability, compliance, mechanism of action and efficacy of QBECO site specific immunomodulation for the induction of clinical response and remission in subjects with moderate to severe ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who have reached age of majority
* Willing to learn and able to self-administer study drug
* Diagnosis of UC established at least 6 months before screening visit, by clinical and endoscopic evidence.
* Currently experiencing moderate to severe active UC defined as a Mayo score of 6-12 (inclusive) at Screening.
* Endoscopic evidence of active mucosal disease, as assessed by flexible sigmoidoscopy, with an Endoscopic Finding Sub-score of ≥2 at Screening.
* Rectal Bleeding Sub-score of ≥1 at Screening.
* Physician's Global Assessment Sub-score of ≥2 at Screening.
* Male/female subjects who agree to practice effective methods of contraception

Exclusion Criteria:

* History of colonic or rectal surgery other than hemorrhoid surgery or appendectomy
* Currently receiving total parenteral nutrition
* Disease limited to ulcerative proctitis
* Diagnosed with Crohn's disease, indeterminate colitis, microscopic colitis or, ischemic or infectious colitis
* Known or suspected hypersensitivity to any component of the product
* Known human immunodeficiency virus (HIV) infection or other immunosuppressive disorder
* Concurrently participating in another study or receiving other experimental or investigational therapies within past 3 months
* Females who are currently pregnant or lactating
* Any history of malignancy. Exceptions may apply for cervical cancer and some forms of skin cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent AEs and clinically significant changes or abnormalities from physical examinations, vital signs and laboratory results (composite) | Day 1 to Week 56
Proportion of subjects in clinical remission | Week 52
  Mayo score ≤ 2 points, with no individual subscore >1

SECONDARY OUTCOMES:
Proportion of subjects in clinical remission | Week 16
  Mayo score ≤ 2 points, with no individual subscore >1
Proportion of subjects with a clinical response | Week 16
  A decrease of the Mayo score from screening of at least 3 points and at least 30%, AND either a decrease from the pre-treatment screening sub-score for rectal bleeding of at least 1 point, OR rectal bleeding sub-score of 0 or 1
Proportion of subjects with a clinical response | Week 52
  A decrease of the Mayo score from screening of at least 3 points and at least 30%, AND either a decrease from the pre-treatment screening sub-score for rectal bleeding of at least 1 point, OR rectal bleeding sub-score of 0 or 1

OTHER OUTCOMES:
Exploratory variables are presence or absence of single nucleotide polymorphisms; changes in immunological biomarkers in blood and colonic tissue; and changes in GI microbiome. (composite) | up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Qu Biologics
Locations (3):
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - GI Research Institute, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario